## N-of-few Study of Pain Perception (NOF)

NCT04664400

Statistical Analysis Plan

8/3/22

## Statistical analysis plan

Our main statistical analysis will be focused on participants' pain ratings following high vs. low cues for each of the conditions (symbolic learning, conditioning, and instructions only). For each condition, we will report the mean and standard deviation across participants test for significant differences in pain ratings following low vs. high cues with paired t tests, using statistical threshold of alpha = 0.05.

For the counterfactual task, we will compare ratings of the same pain stimulus when it is the better vs. the worst alternative, reporting the mean and SD across participants for this difference, and testing for significance with a paired t test.